CLINICAL TRIAL: NCT04614922
Title: Acceptance and Commitment Therapy-based Rehabilitation of Post-concussion Symptoms: a Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy-based Rehabilitation of Post-concussion Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150525
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Post-Concussion Syndrome; Post-Traumatic Headache
Keywords: Acceptance and Commitment Therapy
MeSH Terms: conditions — Post-Concussion Syndrome; Post-Traumatic Headache | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Participation in a 4 week group program based on Acceptance and Commitment Therapy, individual councelling and home lessions.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- control group (No Intervention): Standard care, i.e. follow-up as needed, to some degree dependent on current capacity of therapists.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — ACT-based rehabilitation is an interdisciplinary group rehabilitation which includes 7 sessions of group-based ACT therapy. Each session lasts 2½ hours and is offered twice a week. The ACT sessions will be based on a detailed intervention manual, developed specifically for group treatment. Each group will include a maximum of eight patients. The patients are asked to do homework between each ACT-group session.
  Other Names: ACT
  Arms: Acceptance and Commitment Therapy

SUMMARY:
The investigators aim to evaluate effects of an outpatient rehabilitation program based on Acceptance and Commitment Therapy compared to usual care on function in patients with post-concussion syndrome (PCS) and post-traumatic headache (PTH). This study builds on the investigators' previous observational studies and treatment studies in this patient group.

DETAILED DESCRIPTION:
The study is run in an outpatient setting at the Department of Physical Medicine and Rehabilitation, St. Olavs Hospital, Trondheim University Hospital, Norway. All patients are also participants in the observational study: "Minimal and mild head injury: an exercise and outpatient follow-up study at St. Olavs Hospital" (REK number 2018/2159).

ELIGIBILITY:
Inclusion Criteria:

* Having sustained a minimal HI or MTBI
* PCS/ PTH had evolved within 1 week after the head trauma.
* At least one post-concussion symptoms of at least moderate degree, that affects daily life.
* > 6 months post-injury.
* First line treatment has been tried, e.g. psychoeducation, increase of physical activity and pharmacological treatments for headache

Exclusion Criteria:

* More than 5 years since last injury.
* Symptoms are better explained by other conditions.
* Severe communication problems, typically due to poor knowledge of Norwegian.
* Severe psychiatric, neurological, somatic or substance abuse disorders that will make it problematic to function in a group and/or will complicate follow-up and outcome assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Postcincussion symptom burden | 3, 6 and 12 months after the intervention
  The Rivermead postconcussion symptom questionnaire. The scale measures 13 common postconcussion somatic, emotional and cognitive symptoms on a range from 0 (no symptoms) to 64 (all symptoms graded as severe).

SECONDARY OUTCOMES:
Headache | 3, 6 and 12 months after the intervention
  mean change in days of headache of at least moderate intensity, based on headache diary
Work participation | 3, 6 and 12 months after the intervention
  change in the self-reported number of hours with paid work or ordinary studies per week

OTHER OUTCOMES:
Change of level of cytokines in peripheral blood | at baseline and at 3 months after the intervention
  Blood tests are collected before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Toril Skandsen, phd, Principal Investigator — Norwegian University of Science and Technology, INB; Brit-Elin Lurud, md, Study Director — St. Olavs hospital, Clinic of Rehabilitation
Locations (1):
- St Olavs Hospital Clinic of Physical Medicine and Rehabilitation, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No